CLINICAL TRIAL: NCT07383467
Title: No Time to Wait: A Randomized Control Trial of Online Single-Session Intervention for Children and Adolescents on Psychotherapy Waitlists in Hong Kong
Brief Title: No Time to Wait: Single Session Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Christian Hospital (Other)
Collaborators: Hong Kong University (Other)
Responsible Party: Principal Investigator, Timmy Tsoi, Clinical Psychologist, United Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAED-2025-077
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Anxiety
Keywords: Single Session Intervention; Youth; Depression and Anxiety; Alexithymia
MeSH Terms: conditions — Anxiety Disorders; Depression; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who receive online single session intervention
  Interventions: Other: Online Single Session Intervention on Growth Mindset
- Control Group (No Intervention): Waitlist Control

INTERVENTIONS:
Other: Online Single Session Intervention on Growth Mindset — Participants would receive an online single session intervention, which includes animation and exercises that enhance children and adolescents' growth mindset
  Arms: Intervention Group

SUMMARY:
Mental health problems in youth are prevalent, but early intervention effectively reduces symptoms, substance abuse risk, suicide, and comorbidities. In Hong Kong, however, only 26% of people with common mental disorders seek services (Lam et al., 2015), and even then, they face long delays-e.g., 90 weeks (90th percentile) for stable cases in public psychiatry clinics (Hospital Authority, 2024). Barriers include high costs, transportation issues, stigma, and preference for self-help, creating a strong need for scalable, accessible digital solutions, especially for youth.

Single-Session Interventions (SSI) offer promise as brief, time-efficient tools that provide immediate support with minimal engagement burden. Online SSIs are often free, publicly available, and evidence-based. Research shows they reduce symptoms (moderate effect size Hedges' g = 0.32; 58% chance of better outcome vs. control), improve functioning, and boost satisfaction (Schleider & Weisz, 2017). They work well for specific phobias and acute stress. Yet, their real-world acceptability, effectiveness outside trials, and integration with public services remain understudied-particularly for children/adolescents on waitlists.

This pilot study evaluates an online single-session psychotherapy for youth (children/adolescents) on Hong Kong public psychotherapy waitlists, targeting depression and anxiety symptoms. It extends prior work by:

Targeting two key constructs prominent in Asian contexts:

Alexithymia - difficulty identifying/describing emotions; affects ~10% generally but 36% of Hong Kong adolescents (higher in females). It worsens depression, lowers well-being, complicates therapy, and reduces help-seeking.

Fixed mindset (vs. growth mindset) - Asian groups show lower growth mindset levels; growth mindset buffers mental health issues (meta-analysis r = -0.220 with anxiety/depression/stress) and promotes better emotional regulation and treatment engagement.

Examining how SSI influences acceptability and expectancy toward subsequent face-to-face psychotherapy.

Hypotheses:

SSI will reduce depression/anxiety symptoms more than treatment-as-usual. SSI will increase acceptability and positive expectancy for future in-person treatment.

Change mechanisms-perceived behavioral control and emotional control-will mediate and sustain post-intervention outcomes.

Overall, the study aims to test SSI as a bridge intervention to bridge service gaps, address culturally relevant barriers, and inform scalable mental health strategies in resource-constrained settings like Hong Kong's public system.

DETAILED DESCRIPTION:
Early intervention has been shown to effectively reduce symptoms of mental disorder, and the subsequent risk of substance abuse, suicide, and other mental disorders (Catania et al., 2014; McGorry et al., 2018). However, in Hong Kong, only 26% of individuals with common mental health disorders seek any mental health service (Lam et al., 2015). Even when help is sought, those in need often face lengthy waiting time before receiving treatment, which can have detrimental effects on their mental well-being. For individuals categorized as stable, the average 90th percentile waiting time for psychiatry specialist outpatient clinics amounted to 90 weeks. (Hospital Authority, 2024) Numerous systemic and internal barriers further impede access to mental health services, particularly for youth. These barriers include high costs, transportation challenges, stigma, and a preference for self-help options (Calati & Courtet, 2016; Wampold et al., 2011). As the result, there is a pressing need for scalable and accessible digital interventions that can address the gap in service delivery.

Single-session intervention (SSI) has emerged as a time-efficient and accessible intervention that may provide immediate support and mitigate the negative impact of mental health issues (Campbell, 2012; Schleider & Weisz, 2017). Online SSIs, in particular, hold substantial promise for addressing many challenges associated with traditional digital mental health tools. They can be completed in a single sitting, minimizing user engagement burdens, and many of them are cost-free, publicly accessible, and incorporate evidence-based intervention components. Despite these advantages, the acceptability and effectiveness of online SSIs outside of controlled clinical trials, as well as their synergy with public mental health services, remained underexplored. This study seeks to fill this gap by evaluating the effectiveness and acceptability of single-session psychotherapy for children and adolescents on psychotherapy waitlists in Hong Kong.

Research on SSIs highlights its potential benefits in addressing mental health concerns in a time-limited manner. Single-session interventions, such as the "Walk-in Clinic" and online self-help model, have been implemented successfully in various settings, demonstrating positive outcomes for individuals with a range of psychological difficulties (Rees et al., 2020; Schleider & Weisz, 2017). Studies have shown that single-session interventions can lead to significant symptom reduction, improved functioning, and increased patient satisfaction (Wampold, 2015). A meta-analysis has shown that the calculated effect size (ES) at the end of the intervention was found to be 0.32 according to Hedges' g, indicating a moderate positive impact. This suggests that there was a 58% likelihood of an adolescent who received the single-session intervention (SSI) experiencing better outcomes compared to a youth in the control group (Schleider & Weisz, 2017). Moreover, single-session psychotherapy has been found to be particularly effective for certain conditions, such as specific phobias and acute stress reactions (Rosenbaum et al., 2017; Sloan et al., 2018).

However, limited research has specifically examined the application of single-session psychotherapy for children and adolescents on public mental health service waitlist. Understanding the potential benefits and limitations of single-session psychotherapy in this context can inform mental health service providers and policymakers in developing efficient and accessible interventions for children and adolescents. This study will examine the possibility of SSI in enhancing participants' acceptability toward future psychotherapy. Furthermore, it aims to address specify personality constructs - alexithymia and fixed mindset - that impede the recovery process and are particularly prominent within Asian culture context.

Alexithymia, a condition marked by difficulties in processing emotions and distinguishing them from physical sensations, affects approximately 10% of the general population (Salminen et al., 1999; Samur et al., 2013). However, research indicates that 36% of adolescents in Hong Kong exhibit alexithymic traits, with 34.3% of males and 40% of females affected (Ng & Chan, 2020). First described by Sifneos (1973), alexithymia has been linked in neurobiological studies to impairments in identifying emotions in others (Jongen et al., 2014; Moriguchi & Komaki, 2013). This condition can worsen depressive symptoms (Günther et al., 2016) and diminish overall well-being (Timoney & Holder, 2013). Moreover, alexithymia complicates psychological treatments, often leading to poorer therapeutic outcomes in managing other psychiatric disorders (Ogrodniczuk et al., 2005; Porcelli et al., 2017) and reducing the likelihood of seeking help (Makris, 2023).

In addition to alexithymia, Asian populations tend to exhibit lower levels of growth mindset compared to Western populations (Sun et al., 2021). A growth mindset, which reflects the belief in one's capacity for improvement and development, is recognized as a potential buffer against mental health challenges. Emerging research highlights the positive relationship between growth mindset and mental health. For example, a meta-analysis revealed a moderate negative association (r = -0.220, 95% CI = -0.257, -0.184, p < 0.001) between growth mindset and psychological issues such as anxiety, depression, stress, and low well- being (Burnette et al., 2020). Individuals with a growth mindset are more likely to adopt healthier emotional regulation strategies, including seeking professional support.

Additionally, those with growth mindsets regarding substance addiction demonstrate more favorable attitudes toward treatment (Grand, 2001), while those with growth mindsets about personality are more likely to engage positively with counseling and show greater commitment to therapy (Angilella, 2005).

This pilot study is the empirical study that aims at evaluating the efficacy of an online single session intervention for depression and anxiety symptoms. It will also extend the past research in the following ways: (1) the research will further explore the efficacy and effectiveness of targeting alexithymia and growth mindset in a single session intervention; (2) how single-session intervention affects the treatment expectancy and acceptability of subsequent face-to-face treatment. We hypothesize that (1) the single-session intervention will be more effective in reducing depression and anxiety symptoms compared to a treatment-as-usual group; (2) single-session psychotherapy will enhance the participants' acceptability and expectancy of subsequent face-to-face treatment; (3) mechanisms of change, including perceived primary behavioural control and perceive emotional control, will contribute to and maintain the post- treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

(1) being Hong Kong residents aged 12 - 17; (2) having anxiety and/or depression symptoms, scoring 10 or above, in accordance with Patient Health Questionnaire (PHQ-9) or General Anxiety Disorder-7 (GAD-7); (3) having access to the internet and a valid email address for communication, (4) being able to understand and read Chinese and, (5) participants' parent or legal guardian will be willing to give informed consent.

Exclusion Criteria:

(1) they have received another psychological treatment for depression and/or anxiety in the past 3 months, (2) they report a diagnosis of other comorbid severe psychiatric disorder, including psychotic disorder, bipolar disorder, dissociative disorder, or other neurocognitive disorders that make participation infeasible or interfere with the adherence to the digital self-help intervention, (3) they would participate in another similar study concurrently, (4) any suicidal ideation is reported (score > 2 on Question 9 of the Beck Depression Inventory), (5) they report substance abuse history, (6) having changes in psychotropic medication within 2 weeks before baseline assessment; or (7) they report pregnancy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | From enrolment to 1 month after the end of treatment
GAD-7 | From enrolment to 1 month after the end of treatment
TAS- 20-C | From enrolment to 1 month after the end of treatment
  Alexithymia will be measured using the Toronto Alexithymia Scale (TAS-20), a validated self-report questionnaire assessing difficulty in identifying and describing feelings. The TAS- 20-C is a 20-item self-report scale rated on a five-point Likert scale. It includes three subscales: Difficulty Identifying Feelings (DIF) with items like "When I am upset I don't know if I am sad, frightened, or angry"; Difficulty Describing Feelings (DDF) with statements such as "I find it hard to describe how I feel about people"; and Externally Oriented Thinking (EOT), exemplified by "I prefer to just let things happen rather than to understand why they turned out that way." Scores can range from 20 to 100, where higher scores denote higher alexithymia. The TAS-20-C is validated for Chinese populations (Zhu et al., 2007). In this research, the scale achieved a Cronbach's alpha of 0.80.

SECONDARY OUTCOMES:
Perceived primary (behavioral) control | From Enrolment to 1 month after the end of treatment
  The level of perceived primary control will be evaluated at the beginning, immediately after the intervention, and during the subsequent follow-up using the Perceived Control Scale for Children (PCSC; Weisz, Southam-Gerow, & McCarty, 2001). This scale consists of 24 items that measure the perceived ability to exert primary control, which refers to influencing objective events or conditions through personal effort. Participants will indicate their level of agreement with statements regarding their perceived primary control in the face of social and academic challenges.
Perceived secondary (emotional) control | From enrolment to 1 month after the end of treatment
  Similar to perceived primary control, perceived secondary control will be assessed at baseline, post-intervention, and the follow-up using the Mindset of Depression Anxiety and Stress Scale (MDASS; Zhu et al., 2022). The MDASS is a 12-item scale that measures the perceived capacity for secondary control, which involves influencing the personal psychological impact of objective conditions by adjusting oneself to fit those conditions. Respondents will rate their level of agreement with items reflecting perceived secondary control of various types, such as finding a positive aspect in distressing situations.
Attitudes Toward Seeking Professional Psychological Help (ATSPPH) Short Form | From enrolment to 1-month after the end of treatment
  Acceptability towards professional help is a 10-item questionnaire assessing attitudes towards seeking psychological support. It evaluates participants' recognition of the need for help, stigma tolerance, interpersonal openness, and confidence in mental health practitioners. Items are scored on a four-point Likert scale from 0 to 3, with mean scores calculated for each subscale. This scale has been validated in both Western and Eastern samples (e.g., Hatchett, 2006; Masuda et al., 2005). Previous research has shown it to have strong reliability (α = .86), as supported by this study (α = .79).

CONTACTS AND LOCATIONS:
Locations (1):
- United Christian Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided